CLINICAL TRIAL: NCT03044678
Title: School Based Prevention for Childhood Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Armando Pina, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MH086687
Record Dates: First submitted 2017-01-30; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Masked or blinded to hypotheses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: REACH for Success (Experimental): Experimental: Exposure-based, cognitive and behavioral, social skills training intervention 6-weeks - 6 session -20-30 min each
  Interventions: Behavioral: REACH for Success
- Active Comparator: Self-study (Active Comparator): Active Comparator: Books "What to do when you are scared and worried?How to do homework without throwing-up? How to get organized without losing it?" Reading at home
  Interventions: Behavioral: Self-Study

INTERVENTIONS:
Behavioral: REACH for Success — Exposure-based cognitive behavioral with social skill training (cognitive self control, relaxation, skills for conversations and assertiveness)
  Arms: Experimental: REACH for Success
Behavioral: Self-Study — Books for youth about anxiety management
  Arms: Active Comparator: Self-study

SUMMARY:
This study was designed to conceptualize a school-based prevention program or childhood anxiety.

DETAILED DESCRIPTION:
This is a project corresponding to a career development grant. The main goal of the proposed research was to identify potential barriers to implementing a school-based anxiety preventive intervention, identify strategies to overcome these barriers, and use this information to test a school-based indicated intervention for child anxiety.

ELIGIBILITY:
Inclusion:

Borderline child anxiety levels based on the Spence Child Anxiety Scale

Exclusion:

Externalizing problems (based on teacher nominations) more severe than Spence Child Anxiety Scale borderline levels

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Change in child anxiety symptoms (clinical) | Change from baseline to 12-month follow-up
  Child anxiety symptoms based on the Multidimensional Anxiety Scale for Children
Change in child anxiety levels (typical) | Change from baseline to 12-month follow-up
  Child anxiety based on the Spence Child Anxiety Scale

SECONDARY OUTCOMES:
Changes in child negative cognition | Change from baseline to immediate posttest (at 6-weeks)
  Children's Negative Cognitive Errors on the Children's Negative Cognitive Errors Questionnaire
Changes in child negative cognition | Change from baseline to 12-month follow-up
  Children's Negative Cognitive Errors on the Children's Negative Cognitive Errors Questionnaire
Changes in emotion understanding and expression | Change from baseline to immediate posttest (at 6-weeks)
  Children's Emotion Expressivity based on the Emotion Expressivity Scale for Children
Changes in emotion understanding and expression | Change from baseline to 12-month follow-up)
  Children's Emotion Expressivity based on the Emotion Expressivity Scale for Children
Changes in self efficacy | Change from baseline to immediate posttest (at 6-weeks)
  Child self efficacy based on the Children's Self-Efficacy Questionnaire for Handling School Situations
Changes in self efficacy | Change from baseline to 12-month follow-up)
  Child self efficacy based on the Children's Self-Efficacy Questionnaire for Handling School Situations
Changes in child social skills | Change from baseline to immediate posttest (at 6-weeks)
  Child social skills based on the Social Skills Improvement Rating System
Changes in child social skills | Change from baseline to 12-month follow-up)
  Child social skills based on the Social Skills Improvement Rating System
Changes in somatic arousal | Change from baseline to immediate posttest (at 6-weeks)
  Child somatic arousal based on the Physiological Hyperarousal Scale for Children
Changes in somatic arousal | Change from baseline to 12-month follow-up)
  Child somatic arousal based on the Physiological Hyperarousal Scale for Children

IPD SHARING:
Plan to Share IPD: No